CLINICAL TRIAL: NCT06204120
Title: A Multicenter, Randomized, Double-blind, Placebo, Positive Drug Parallel Controlled Phase II Clinical Trial to Evaluate the Efficacy and Safety of LPM3480392 Injection for Moderate to Severe Pain After Abdominal Surgery
Brief Title: Phase II Clinical Trial to Evaluate the Efficacy and Safety of LPM3480392 Injection for Moderate to Severe Pain After Abdominal Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LY03014/CT-CHN-203
Record Dates: First submitted 2023-04-22; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- morphine hydrochloride injection (Active Comparator)
  Interventions: Drug: morphine hydrochloride injection
- LPM3480392 injection group 1 (Experimental)
  Interventions: Drug: LPM3480392 Injection
- LPM3480392 injection group 2 (Experimental)
  Interventions: Drug: LPM3480392 Injection
- LPM3480392 injection group 3 (Experimental)
  Interventions: Drug: LPM3480392 Injection
- LPM3480392 injection group 4 (Experimental)
  Interventions: Drug: LPM3480392 Injection

INTERVENTIONS:
Drug: LPM3480392 Injection — PCA administration
  Arms: LPM3480392 injection group 1; LPM3480392 injection group 2; LPM3480392 injection group 3; LPM3480392 injection group 4
Drug: Placebo — PCA administration
  Arms: Placebo
Drug: morphine hydrochloride injection — PCA administration
  Arms: morphine hydrochloride injection

SUMMARY:
A randomized, double-blind, placebo/positive drug parallel controlled design was used to evaluate the preliminary efficacy and safety of intravenous infusion of LPM3480392 injection using different dosing regimens in subjects with moderate to severe pain after abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signed informed consent form (ICF) and comply with the trial procedures before starting the trial-related activities;
2. Aged 18-65 years (including the boundary value), male or female;
3. Body mass index (BMI) 18-29 kg/m2 (including the boundary value), male body weight ≥ 50 kg; female body weight ≥ 45 kg;
4. Subjects scheduled for elective abdominal surgery under general anesthesia, 1h ≤ duration of estimated surgery Interval ≤ 4h;
5. American Society of Anesthesiologists（ASA ）grade I ~ II;
6. Female subjects (not surgically sterile, surgical sterilization is defined as hysterectomy or oophorectomy) with a negative pregnancy test at Screening. Male and female subjects agree to take effective contraceptive measures throughout the study and for at least 1 month after medication;
7. The investigator judges that the patient has recovered from intraoperative anesthesia to enough awake, which can be accurately completed the questionnaire was specified, and the numerical rating scale（NRS） score at rest was ≥ 4 points within 4 hours after surgery.

Exclusion Criteria:

1. Known history of allergy to any component of the investigational product, or allergy or contraindication to the anesthetic/analgesic drugs used in the study;
2. Had any of the following conditions or medical history:

   1. History of stroke, cognitive dysfunction, or epilepsy (excluding convulsions caused by previous febrile convulsions in children);
   2. History of difficult airway, such as obstructive sleep apnea syndrome, bronchial asthma, chronic respiratory diseases or other serious respiratory diseases;
   3. Subjects with a history of myocardial infarction, angina pectoris, severe arrhythmia of degree II or above atrioventricular block, or New York Heart Association（NYHA） Class II or above within 6 months prior to screening;
   4. History of vestibular dysfunction or motion sickness;
   5. Have a history of diabetes and glycosylated hemoglobin ≥ 9% during the screening period;
   6. Esophagitis;
   7. Paralytic gastrointestinal obstruction;
   8. The presence of other acute and chronic pain conditions preoperatively or in combination with other bodily pain conditions that confound the evaluation of postoperative pain.
3. Medications affecting postoperative analgesia before randomization:

   a) Opioid analgesics taken continuously for more than 10 days for any reason within 3 months prior to randomization, or taking opioid analgesics within 7 days prior to randomization; b） Use of the following drugs within 14 days prior to randomization, including but not limited to: ketamine, non-steroidal anti-inflammatory drugs (aspirin, acetaminophen, indomethacin, diclofenac, ibuprofen, parecoxib sodium, etc.), alpha adrenoceptor agonists (dexmedetomidine hydrochloride, clonidine, etc.), glucocorticoids (dexamethasone hydrochloride, hydrocortisone, methylprednisolone, etc., except for topical or topical use of glucocorticoids), antiepileptic drugs (carbamazepine, sodium valproate, etc.), sedative drugs (diazepam, estazolam, midazolam, alprazolam, barbiturate, phenobarbital and chloral hydrate, etc.); c） Use of Chinese herbal medicine or Chinese patent medicine within 7 days prior to randomization.
4. Systolic blood pressure less than 90 mmHg or greater than 160 mmHg and diastolic blood pressure less than 1 day before surgery 60 mmHg or greater;
5. Peripheral saturation (SpO2) < 92% at screening or before administration;
6. corrected QT interval（QTc ）> 450 ms for males and > 460 m for females at screening or pre-dose ( QTc is expressed as Fridericia formula calculation);
7. Patients with abnormal liver and kidney function during screening period or before administration: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) > 1.5 times of normal value, total bilirubin higher than the upper limit of normal value, serum creatinine (Cr) > 1.5 times of the upper limit of normal value during screening period;
8. Subjects with coagulation abnormalities (PT prolonged more than 3 seconds above the upper limit of normal and/or activated partial thromboplastin time（APTT） prolonged more than 10 seconds above the upper limit of normal) during the screening period; and the investigator confirmed that the abnormalities were clinically significant;
9. History of drug abuse or drug abuse before screening;
10. Positive result in screening of drugs of abuse via urinalysis;
11. Nursing mothers;
12. Positive hepatitis B virus surface antigen (HBsAg) test [but the subject is eligible if the peripheral blood hepatitis B virus deoxyribonucleic acid (HBV DNA) is lower than the lower limit of the reference range, and the investigator believes that the subject is in a stable phase of chronic hepatitis B and will not increase the risk of the subject]; hepatitis C virus (HCV) antibody, treponema pallidum antibody, human immunodeficiency virus (HIV) antibody positive;
13. Participation in any medication (excluding vitamins and minerals) within 3 months prior to informed consent Quality) Clinical trial personnel, except for those not using investigational drugs;
14. subjects who are judged by the investigator to be not suitable for this clinical trial, including but not limited to the presence of conditions that may confound the interpretation of efficacy, safety, or tolerability data in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-11-25 (Actual); Primary Completion 2023-07-04 (Actual); Study Completion 2023-07-04 (Actual)

PRIMARY OUTCOMES:
SPID24(the Sum of Pain Intensity Differences in Pain Score from baseline Over 24 Hours) | one day
  Pain intensity will be evaluated using an 11-point (0-10) Numeric Pain Rating Scale (NPRS), with higher numbers indicating a higher pain intensity, administered over 24 hours.

SECONDARY OUTCOMES:
Cumulative dose of rescue analgesic drugs within 24 h | one day
Percentage of subjects not using rescue analgesic medication within 24 h | one day
Time of the first rescue analgesic drug | one day
Total number of compressions within 24 hours. | one day
Incidence and severity of adverse events within 24 h | one day
Sedation scale score | one day
Respiratory depression events (defined as respiratory rate ≤ 8 breaths/min and/or saturation < 90%) | one day

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital Affiliated to Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No